CLINICAL TRIAL: NCT06181799
Title: Biomarkers of the Exhaled Breath and Single-Lead Electrocardiography in the Diagnosis of Myocardial Ischemia
Brief Title: Volatilome and Single-Lead Electrocardiogram Optimize Ischemic Heart Disease Diagnosis Using Machine Learning Models
Status: Completed | Type: Observational
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 13011998
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2023-10

CONDITIONS: Coronary Artery Disease; Ischemic Heart Disease; Chronic Coronary Disease; Angina Pectoris; Stable Coronary Artery Disease CAD
Keywords: Coronary Artery Disease; Mass Spectrometry; Volatilome; Single Lead-ECG; Ischemic Heart Disease; Lipidome; Inflammasome; Electrocardiography; PTR-TOF-MS-1000; Stress Induced Myocardial Perfusion Defect; Qardio-Qvark; Stable Coronary Artery Disease; Atherosclerosis; Breathome; Volatile Organic Compound; Bicycle Ergometry; Prevention; SCORE2; SCORE2-OP; Smart Risk Score; Machine Learning Model; Artificial intelligence; Cardiovascular disease; Risk Factor; Angina pectoris
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Angina Pectoris; Atherosclerosis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: The group is planned to include 31 people with myocardial perfusion defect on the stress computed tomography myocardial perfusion Imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Interventions: Diagnostic Test: Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).
- Control group: The group is planned to include 49 people without myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Interventions: Diagnostic Test: Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).

INTERVENTIONS:
Diagnostic Test: Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe). — Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models.

SUMMARY:
This is a prospective, case-control, single-center, observational, non-randomized study. It is designed to evaluate the diagnostic accuracy of functional tests involving physical exertion monitored via a 12-lead ECG, combined with analysis of exhaled breath volatile organic compounds (VOCs) and single-lead ECG parameters.

DETAILED DESCRIPTION:
The planned number of participants to include in the study is 80, admitted to the University Clinical Hospitals No. 1, at the I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University).

The study includes the following stages:

1. Participants will be selected according to inclusion and exclusion criteria;
2. Work with medical documentation;
3. Instrumental and laboratory examinations of the participants:

3.1. Analysis of exhaled air will be carried out with the Compact PTR-MS instrument manufactured by Ionicon (Austria) (analytical device), registration certificate No. (C16)07/C05.

3.2. All the participants will undergo a single blood sampling during the day of performing the study, a blood test, 10 ml from a peripheral vein to determine the level of total cholesterol, low-density lipoprotein (LDL), very low-density lipoprotein (VLDL), high-density lipoprotein (HDL), triglycerides, C-reactive protein (CRP), lipoprotein a, apolipoprotein B, and interleukin-6 (IL-6).

3.3. Both groups will perform a bicycle ergometry test (on a SCHILLER c200 device) to evaluate the response to physical activity.

3.4. Before and immediately after the exercise test, all patients are scheduled to record a single-lead ECG and pulse wave, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow).

4.5. Stress computed tomography myocardial perfusion imaging (CTP) with a vasodilation test using adenosine triphosphate on a CT device with 640 slices (Canon; Aquilion One Genesis) will be performed.

After completion of the instrumental and laboratory analysis, a statistical analysis will be conducted using classical statistics and machine learning methods, including gradient boosting.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥40 years;
2. Absence of acute exacerbations of psychiatric disorders or cognitive impairments that would preclude study participation;
3. Provision of written informed consent for study participation, blood sample collection, and anonymous publication of research results;
4. Pre-test probability of ischemic heart disease between 1% and 33%.

Non-inclusion criteria:

1. Pregnancy and breastfeeding;
2. Diabetes mellitus;
3. Presence of acute myocardial ischemia (acute coronary syndrome or myocardial infarction within the preceding 48 hours) or a history of myocardial infarction;
4. Active infectious or non-infectious inflammatory diseases in the acute/exacerbation phase;
5. Connective tissue diseases (regardless of disease activity);
6. Respiratory disorders (e.g., bronchial asthma, chronic bronchitis, cystic fibrosis, or other conditions associated with significant respiratory dysfunction);
7. Acute pulmonary thromboembolism involving the pulmonary artery or its branches;
8. Aortic dissection;
9. Hemodynamically significant decompensated cardiac valvular defects**;
10. Active malignancy;
11. Decompensated chronic heart failure (NYHA class III-IV) or acute heart failure;
12. Neurological disorders (e.g., Parkinson's disease, multiple sclerosis, acute psychosis, Guillain-Barré syndrome);
13. Cardiac arrhythmias or conduction abnormalities contraindicating stress testing;
14. Musculoskeletal disorders precluding exercise testing (e.g., bicycle ergometry);
15. Allergy to radiocontrast agents and/or adenosine triphosphate (ATP);
16. Chronic kidney disease with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m² (CKD-EPI formula);
17. Severe hepatic insufficiency and/or Child-Pugh class B or C liver cirrhosis.

Exclusion Criteria:

1. Poor recording quality of single-channel electrocardiogram (ECG) and/or plethysmography data;
2. Failure to complete the stress test due to reasons unrelated to cardiac conditions;
3. Voluntary withdrawal of consent to continue participation in the study;
4. Post-enrollment development of conditions or identification of pathologies listed in the exclusion criteria.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The planned number of participants to include in the study is 80, admitted to the University Clinical Hospitals No. 1, at the I.M. Sechenov First Moscow State Medical University of the Ministry of Health of the Russian Federation (Sechenov University).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Kopylov, Professor, Principal Investigator — I.M. Sechenov First Moscow State Medical University (Sechenov University)
Locations (1):
- Federal State Budgetary Educational Institution of Higher Education First Moscow State Medical University named after I.M. Sechenov of the Ministry of Health of Russia, City Clinical Hospital No. 1, Cardiology Clinic, Institute of Personalized Cardiology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No
No, due to the prohibition by the local ethical committee

REFERENCES:
- [Background] Marzoog BA, Kopylov P. Volatilome and machine learning in ischemic heart disease: Current challenges and future perspectives. World J Cardiol. 2025 Apr 26;17(4):106593. doi: 10.4330/wjc.v17.i4.106593. PMID 40308617
- [Background] Marzoog BA, Chomakhidze P, Gognieva D, Parunova AY, Demchuk SN, Silantyev A, Kuznetsova N, Kostikova A, Podgalo D, Nagornov E, Gadzhiakhmedova A, Kopylov P. Updates in breathomics behavior in ischemic heart disease and heart failure, mass-spectrometry. World J Cardiol. 2025 Feb 26;17(2):102851. doi: 10.4330/wjc.v17.i2.102851. PMID 40061284
- [Background] Marzoog B. Breathomics Detect the Cardiovascular Disease: Delusion or Dilution of the Metabolomic Signature. Curr Cardiol Rev. 2024;20(4):e020224226647. doi: 10.2174/011573403X283768240124065853. PMID 38318837
- [Background] Marzoog BA, Gognieva D, Chomakhidze P, Kopylov P. Cardi-Ankle Vascular Index Optimizes Ischemic Heart disease Diagnosis. MedRxiv 2024:2024.07.03.24309877. https://doi.org/10.1101/2024.07.03.24309877.
- [Background] Marzoog BA. Volatilome: A Novel Tool for Risk Scoring in Ischemic Heart Disease. Curr Cardiol Rev. 2024;20(6):e080724231719. doi: 10.2174/011573403X304090240705063536. PMID 38982923
- [Background] Marzoog BA. Volatilome is Inflammasome- and Lipidome-dependent in Ischemic Heart Disease. Curr Cardiol Rev. 2024;20(6):e190724232038. doi: 10.2174/011573403X302934240715113647. PMID 39039680
- [Result] Marzoog BA, Chomakhidze P, Gognieva D, Silantyev A, Suvorov A, Abdullaev M, Mozzhukhina N, Filippova DA, Kostin SV, Kolpashnikova M, Ershova N, Ushakov N, Mesitskaya D, Kopylov P. Development and validation of a machine learning model for diagnosis of ischemic heart disease using single-lead electrocardiogram parameters. World J Cardiol. 2025 Apr 26;17(4):104396. doi: 10.4330/wjc.v17.i4.104396. PMID 40308623
- [Result] Marzoog BA, Abdullaev M, Suvorov A, Chomakhidze P, Gognieva D, Gagarina NV, et al. Single Channel Electrocardiography Optimizes the Diagnostic Accuracy of Bicycle Ergometry! MedRxiv 2024:2024.04.20.24306122. https://doi.org/10.1101/2024.04.20.24306122.
- [Result] Marzoog BA, Chomakhidze P, Kopylov P. Reevaluation of the Bicycle Ergometry in the Diagnosis of Ischemic Heart Disease. MedRxiv 2024:2024.07.03.24309879. https://doi.org/10.1101/2024.07.03.24309879.
- [Result] B.A. Marzoog, P. Chomakhidze, A. Suvorov, P. Kopylov, CARDIO-QVARK Diagnose Ischemic Myocardiocyte!, (n.d.). https://doi.org/10.1101/2024.07.16.24310485.
- [Result] Marzoog BA, Chomakhidze P, Gognieva D, Gagarina NV, Silantyev A, Suvorov A, Fominykha E, Mustafina M, Natalya E, Gadzhiakhmedova A, Kopylov P. Machine Learning Model Discriminate Ischemic Heart Disease Using Breathome Analysis. Biomedicines. 2024 Dec 11;12(12):2814. doi: 10.3390/biomedicines12122814. PMID 39767720
- [Result] Marzoog BA, Chomakhidze P, Gognieva D, Silantyev A, Suvorov A, Stroeva A, Mustafina M, Fedorova AY, Syrkin A, Kopylov P. Exhaled Breath Biomarkers Reflect the Inflammasome and Lipidome Changes in Ischemic Heart Disease: A Study Using Machine Learning Models and Network Analysis. J Lipid Atheroscler. 2025 Sep;14(3):350-371. doi: 10.12997/jla.2025.14.3.350. Epub 2025 Jul 8. PMID 41048598

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Group: The group is planned to include 31 people with myocardial perfusion defect on the stress computed tomography myocardial perfusion Imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).: Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models.
- Control Group: The group is planned to include 49 people without myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).: Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models.
Period: Overall Study
Arm/Group | Experimental Group | Control Group
Started | 31 | 49
Completed | 31 | 49
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group | Control Group | Total
Number analyzed (Participants) | 31 | 49 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] — The patients were collected from the Sechenov University clinical hospital number 1
  years | 59.93 (11.70) | 53.96 (9.23) | 56.28 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 22 | 39
  Male | 14 | 27 | 41
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 31 | 49 | 80

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy (AUC, Sensitivity, Specificity, NPV, PPV) of the Stress-ECG Test in Ischemic Heart Disease
Description: Assessing the diagnostic accuracy of the stress electrocardiography test in ischemic heart disease
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 6 months for the stress electrocardiography test
Measure: Number (95% Confidence Interval); unit: Proportion probability
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
Proportion probability
  AUC | 0.507 [0.388 to 0.625] | 0.507 [0.388 to 0.625]
  Sensitivity | 0.484 [0.306 to 0.657] | 0.484 [0.306 to 0.657]
  Specificity | 0.531 [0.392 to 0.673] | 0.531 [0.392 to 0.673]
  NPV NPV NPV NPV | 0.619 [0.465 to 0.758] | 0.619 [0.465 to 0.758]
  PPV | 0.395 [0.238 to 0.553] | 0.395 [0.238 to 0.553]

2. Primary Outcome: Diagnostic Accuracy (AUC, Sensitivity, Specificity, NPV, PPV) of Exhaled Breath Analysis for Ischemic Heart Disease
Description: Analyze the volatile organic compounds of the exhaled breath in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test (adenosine triphosphate) and compare them with individuals without stress-induced myocardial perfusion defect after a physical stress test, and compare them with rest results as independent variables. Machine learning model was used to assess the diagnostic accuracy of the exhaled breath in the diagnosis of ischemic heart disease
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 6 months for the obtained volatilome data.
Measure: Number (95% Confidence Interval); unit: Proportion probability
Groups:
- Experimental Group: The group includes 31 people with stress-induced myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) with adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)) during 1 minute. Machine learning model is employed to analyze the patterns identified in the exhaled air volatilome data.
  The assessed predictors exceed 750 because the participants exhaled three times at each time. The method used to evaluate these results is calculating delta and then selecting the 5 or 10 most mathematically important predictors for the diagnosis of positive stress-induced myocardial perfusion defect using the machine learning model. Then building the final machine learning model and checking its features, AUC, sensitivity, specificity, PPV, and NPV. For full results check the paper DOI: 10.3390/biomedicines12122814
- Control Group: The group includes 49 people without stress-induced myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) with adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)) during 1 minute. Machine learning model is employed to analyze the patterns identified in the exhaled air volatilome data.
  The assessed predictors exceed 750 because the participants exhaled three times at each time. The method used to evaluate these results is calculating delta and then selecting the 5 or 10 most mathematically important predictors for the diagnosis of positive stress-induced myocardial perfusion defect using the machine learning model. Then building the final machine learning model and checking its features, AUC, sensitivity, specificity, PPV, and NPV. For full results check the paper DOI: 10.3390/biomedicines12122814
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
Proportion probability
  AUC | 0.838 [0.736 to 0.914] | 0.838 [0.736 to 0.914]
  Sensitivity | 0.839 [0.692 to 0.964] | 0.839 [0.692 to 0.964]
  Specificity | 0.776 [0.666 to 0.889] | 0.776 [0.666 to 0.889]
  NPV | 0.884 [0.771 to 0.975] | 0.884 [0.771 to 0.975]
  PPV | 0.703 [0.559 to 0.849] | 0.703 [0.559 to 0.849]

3. Primary Outcome: Diagnostic Accuracy (AUC, Sensitivity, Specificity, NPV, PPV) of Single-Lead ECG With Pulse Wave Analysis in Ischemic Heart Disease
Description: Analyze the parameters of the single-lead electrocardiogram with pulse wave function in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test and compare them with individuals without stress-induced myocardial perfusion defect as an independent variable. Machine learning model was used to assess the diagnostic accuracy of the single-lead ECG with pulse wave function in the diagnosis of ischemic heart disease.
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 6 months for the single lead ECG parameters with pulse wave function
Measure: Number (95% Confidence Interval); unit: Proportion probability
Groups:
- Experimental Group: The group is planned to include 31 people with myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)): Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.4330/wjc.v17.i4.104396
- Control Group: The group is planned to include 49 people without myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)): Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.4330/wjc.v17.i4.104396
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
Proportion probability
  AUC | 0.67 [0.530 to 0.801] | 0.67 [0.530 to 0.801]
  Sensitivity | 0.516 [0.333 to 0.695] | 0.516 [0.333 to 0.695]
  Specificity | 0.755 [0.628 to 0.880] | 0.755 [0.628 to 0.880]
  NPV | 0.712 [0.586 to 0.830] | 0.712 [0.586 to 0.830]
  PPV | 0.571 [0.387 to 0.758] | 0.571 [0.387 to 0.758]

4. Primary Outcome: Changes in the Concentration of Total Cholesterol, TG (mmol/L), LDL (mmol/L), LDL (mmol/L), HDL (mmol/L), and VLDL (mmol/L) in Individuals With Stress-induced Myocardial Perfusion Defect vs. Without.
Description: Analyzing the taken blood samples for total cholesterol, TG (mmol/L), LDL (mmol/L), LDL (mmol/L), HDL (mmol/L), and VLDL (mmol/L) in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test and comparing them with individuals without stress-induced myocardial perfusion defect as independent variables.
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 1 week for the total cholesterol, TG (mmol/L), LDL (mmol/L), LDL (mmol/L), HDL (mmol/L), and VLDL (mmol/L) data.
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Experimental Group: The group is planned to include 31 people with myocardial perfusion defect on the stress computed tomography myocardial perfusion Imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).: Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.12997/jla.2025.14.e30
- Control Group: The group is planned to include 49 people without myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe).: Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.12997/jla.2025.14.e30
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
mmol/L
  Total cholesterol (mmol/L) | 5.61 (1.56) | 5.49 (1.43)
  TG (mmol/L) | 1.41 (0.77) | 1.16 (0.54)
  LDL (mmol/L) | 3.46 (1.08) | 3.27 (0.96)
  HDL (mmol/L) | 1.28 (0.34) | 1.44 (0.50)
  VLDL (mmol/L) | 0.64 (0.35) | 0.52 (0.25)

5. Primary Outcome: Changes in the Concentration of Apolipoprotein B (g/L) in Individuals With Stress-induced Myocardial Perfusion Defect vs. Without.
Description: Analyzing the taken blood samples for Apolipoprotein B (g/L) in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test and comparing them with individuals without stress-induced myocardial perfusion defect as independent variables.
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 1 week for the Apolipoprotein В (g/L) data.
Measure: Mean (Standard Deviation); unit: g/L
Groups:
- Experimental Group: The group is planned to include 31 people with myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)): Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.12997/jla.2025.14.e30
- Control Group: The group is planned to include 49 people without myocardial perfusion defect on the stress computed tomography myocardial perfusion imaging (by using contrast-enhanced multi-slice spiral computed tomography (CE-MSCT) using adenosine triphosphate (ATP)).
  Mass spectrometry using the PTR TOF-1000 (IONICON PTR-TOF-MS - Trace VOC Analyzer, Eduard-Bodem-Gasse 3, 6020 Innsbruck, Austria (Europe)): Once enrolled in the study, all participants are scheduled to undergo the following tests:
  Analysis of the exhaled breath volatile organic compounds using real-time analytical methods (PTR-TOF-MS-1000; real-time mass spectrometer with ionization by the proton transfer method) before and after the physical exertion test, during 1 minute. Machine learning models will be employed to analyze the patterns identified in the exhaled air volatilome data.
  Before and immediately after the physical exertion test, all participants are scheduled to record a single-lead ECG and pulse wave for 3 minutes, using a portable single-lead recorder (Cardio-Qvark) (Russia, Moscow). Single-lead ECG and pulse wave parameters will be analyzed using machine learning models. For full results check the paper DOI: 10.12997/jla.2025.14.e30
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
g/L | 1.19 (0.35) | 1.08 (0.27)

6. Primary Outcome: Changes in the Concentration of Lipoprotein (а) (mg/L) and c-RP (mg/L) in Individuals With Stress-induced Myocardial Perfusion Defect vs. Without.
Description: Analyzing the taken blood samples for lipoprotein (a) (mg/L) and C-RP (mg/L) in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test and comparing them with individuals without stress-induced myocardial perfusion defect as independent variables.
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 1 week for the lipoprotein (а) (mg/L) and c-RP (mg/L) data.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
mg/L
  lipoprotein (а) (mg/L) | 213.22 (207.23) | 253.67 (252.70)
  c-RP (mg/L) | 3.81 (2.96) | 3.09 (3.33)

7. Primary Outcome: Changes in the Concentration of IL- 6 (pg/mL) in Individuals With Stress-induced Myocardial Perfusion Defect vs. Without.
Description: Analyzing the taken blood samples for IL-6 (pg/mL) in individuals with stress-induced myocardial perfusion defect on stress computed tomography myocardial perfusion imaging (CTP) with vasodilation test and comparing them with individuals without stress-induced myocardial perfusion defect as independent variables.
Time Frame: The study was completed on 10.06.2024; the outcome measure was assessed during 1 week for the IL- 6 (pg/mL) data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Experimental Group | Control Group
Number analyzed (Participants) | 31 | 49
pg/mL | 0.88 (0.91) | 0.86 (1.12)

ADVERSE EVENTS:
Time Frame: Over 1 month
Description: All the adverse events, including the "All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were assesed.
Arm/Group | Experimental Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/49
Other Adverse Events (participants affected / at risk) | 0/31 | 0/49

LIMITATIONS AND CAVEATS:
Breath analysis for CAD diagnosis has limitations: bulky/expensive spirometers need portable VOC-specific devices; small sample size requires larger validation trials for combined ECG-breath biomarkers; lack of standardized protocols/reference databases hinders reproducibility. Statistical bias was mitigated via resampling, normalization, and median statistics. Partial consistency with known physiological patterns supports validity despite constraints.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT06181799/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT06181799/SAP_001.pdf